CLINICAL TRIAL: NCT02465203
Title: A Multi-centre 3-year Follow-up Study to Assess the Viral Activity in Patients Who Failed to Achieve Sustained Virologic Response in Novartis-sponsored Alisporivir-studies for Chronic Hepatitis C Patients
Brief Title: 3-year Follow-up Study to Assess the Viral Activity in Hepatitis C Patients Who Failed Feeder DEB025/Alisporivir Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was prematurely terminated.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CDEB025A2313; 2011-006132-24
Record Dates: First submitted 2015-03-17; First posted 2015-06-08 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-12

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Follow up from feeder studies (Other): Follow up arm
  Interventions: Drug: Previous treatment in DEB025 study

INTERVENTIONS:
Drug: Previous treatment in DEB025 study — Follow-up after DEB025 active study
  Other Names: Data was not collected

SUMMARY:
Follow-up for viral activity, changes in liver function and safety in patients with no SVR24 in feeder studies

DETAILED DESCRIPTION:
The purpose of this study was to follow patients from the feeder studies who have not achieved SVR24 to assess their viral activity, and to assess the changes in liver function and disease, and post-treatment safety over time.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥18
2. Have previously completed a Novartis-sponsored hepatitis C study and received alisporivir or a direct antiviral agent (DAA)
3. Have not achieved SVR24

Exclusion Criteria:

1. Use of any investigational drugs within 5 half-lives of enrollment, or within 30 days of that medication, whichever is longer.
2. Previous use of any course of hepatitis C therapy since the end of the Novartis-sponsored hepatitis C study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-09-06 (Actual); Primary Completion 2014-01-23 (Actual); Study Completion 2014-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (38):
- United States (7):
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Ventura, California
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
- Novartis Investigative Site, Westmead, New South Wales, Australia
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Torono, Ontario, Canada
- Germany (6):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kiel
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Mumbai, Maharashtra, India
- Italy (4):
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
- Poland (2):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, San Juan, Puerto Rico
- Romania (4):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Bucharest, District 3
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Iași
- South Korea (2):
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Pusan
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Taiwan (4):
  - Novartis Investigative Site, Douliu
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Linkou District
  - Novartis Investigative Site, Taichung
- Novartis Investigative Site, Songkhla, Thailand
- Novartis Investigative Site, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
terminated

RESULTS

PARTICIPANT FLOW:
Groups:
- From Study 2210 (N=56): Follow up from feeder study NCT01183169
- From Study 2301 (N=36): Follow up from withdrawn feeder study NCT01318694
- From Study 2211 - Overall (N=13): Follow up from feeder study NCT01215643
Period: Overall Study
Arm/Group | From Study 2210 (N=56) | From Study 2301 (N=36) | From Study 2211 - Overall (N=13)
Started | 56 | 36 | 13
Completed | 0 | 0 | 0
Not Completed | 56 | 36 | 13
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Study terminated by sponsor | 50 | 34 | 11
Not completed — New therapy for study indication | 4 | 0 | 0
Not completed — Patient/guardian decision | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Study 2211 - Overall (N=13): Follow up from feeder study NCT01215643
- Total: Total of all reporting groups
Arm/Group | From Study 2210 (N=56) | From Study 2301 (N=36) | Study 2211 - Overall (N=13) | Total
Number analyzed (Participants) | 56 | 36 | 13 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (9.86) | 53.8 (10.57) | 46.5 (7.88) | 52.3 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 4 | 49
  Male | 33 | 14 | 9 | 56
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 40 | 24 | 6 | 70
  Black | 3 | 0 | 1 | 4
  Asian | 12 | 12 | 6 | 30
  Native American | 0 | 0 | 0 | 0
  Pacific Islander | 0 | 0 | 0 | 0
  Other | 1 | 0 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 26.35 (3.76) | 25.54 (4.08) | 26.24 (4.12) | 26.06 (3.89)
Baseline HCV RNA Load (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 6.32 (1.3375) | 6.19 (0.5171) | 6.17 (1.1974) | 6.26 (1.0959)

OUTCOME MEASURES:

1. Primary Outcome: HCV RNA Sequencing
Description: Persistence of resistance associated variants
Time Frame: 27 months
Population: There was no hypothesis testing in this study, as the study was prematurely terminated.
  4 patients with resistance associated variants have been identified at study start. Study was not powered for 105 participants
Measure: Number; unit: Number of particiants
Groups:
- All Arms: All participants in study
Arm/Group | All Arms
Number analyzed (Participants) | 105
Number of particiants | 4

2. Secondary Outcome: Safety Parameters as Measured by HCV RNA Sequencing
Description: Phenotypic analysis of HCV isolates to determine the patients susceptibility/resistance to alisporivir in vitro
Time Frame: 27 months
Population: There was no hypothesis testing in this study, as the study was prematurely terminated.
  Study was powered for efficacy of 650 participants, and only 105 were randomized
  No data are available because data were not collected
Arm/Group | All Arms
Number analyzed (Participants) | 0

3. Secondary Outcome: Safety Parameters as Measured by FibroScan/Fibrotest and Lab Parameters
Description: Changes in liver function and disease over time
Time Frame: 27 months
Population: There was no hypothesis testing in this study, as the study was prematurely terminated.
  No data for any pre-specified Outcomes were analyzed.
  There was no hypothesis testing in this study, as the study was prematurely terminated.
  Study was powered for 105 participants, not 650
  No data are available because data were not collected
Arm/Group | All Arms
Number analyzed (Participants) | 0

4. Secondary Outcome: Safety Parameters as Measured by Liver UltraSound and Lab Parameters
Description: Development of hepatocellular carcinoma (HCC)
Time Frame: 27 months
Population: as for outcome 3
Arm/Group | All Arms
Number analyzed (Participants) | 0

5. Secondary Outcome: Safety Parameters
Description: Safety over time of previous alisporivir exposure
Time Frame: 27 months
Population: There was no hypothesis testing as the study was prematurely terminated. AE and SAE data are provided in the "Adverse Events" section
  There was no hypothesis testing in this study, as the study was prematurely terminated.
  Study was powered for 105 participants, not 650
  No data are available because data were not collected
Arm/Group | All Arms
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- A2210: From Study A2210 (3 patients did not receive alisporivir in the feeder study and were excluded from Safety Set)
- A2301: From Study A2301 (3 patients did not receive alisporivir in the feeder study and were excluded from Safety Set)
- A2211 IFN-free: From Study A2211 IFN-free (subset of Study 2211 overall)
- A2211 Overall: From Study A2211 Overall (1 patient did not receive alisporivir in the feeder study and was excluded from Safety Set)
Arm/Group | A2210 | A2301 | A2211 IFN-free | A2211 Overall
Serious Adverse Events (participants affected / at risk) | 3/53 | 0/33 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 1/53 | 1/33 | 2/6 | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A2210 (N=53) | A2301 (N=33) | A2211 IFN-free (N=6) | A2211 Overall (N=12)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A2210 (N=53) | A2301 (N=33) | A2211 IFN-free (N=6) | A2211 Overall (N=12)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 | 1 | 1 | 2
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 0 | 0 | 0 | 1
TOTAL BILE ACIDS INCREASED (Investigations) | 0 | 0 | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
There is no statistical hypothesis for this single-arm uncontrolled terminated study. Study was powered for efficacy of 650 participants and only 105 were randomized

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Publications from a single site are postponed until publication of the pooled clinical trial data (i.e., data from all sites) or disclosure of trial results in their entirety.